CLINICAL TRIAL: NCT01658111
Title: Robot-aided Therapy in Acute Stroke Patients for the Upper Limb Rehabilitation With Long-term Follow-up.
Brief Title: Robot-aided Therapy in Stroke Patients for Upper Limb Rehabilitation
Acronym: MITEEG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIT02012EEG
Record Dates: First submitted 2012-07-24; First posted 2012-08-06 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2012-08

CONDITIONS: Stroke
Keywords: Stroke; Robots; EEG; EMG
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional physiotherapy (Active Comparator): Each subject will receive 4 weeks of traditional upper limb rehabilitation treatment (20 sessions, 5 days a week for 4 weeks).
  Interventions: Procedure: Traditional physiotherapy
- Robot Group (Experimental): Each subject will be asked to perform five sessions per week goal-directed, planar reaching tasks, which emphasizes shoulder and elbow movements, moving from the centre target to each of 8 peripheral targets equally spaced on a 0.14 m radius circumference around a centre target using the InMotion2 (IM2) system (20 sessions- 5 days a week for 4 weeks).
  Interventions: Device: Robot Group

INTERVENTIONS:
Device: Robot Group — The MIT-MANUS/InMotion2 (Interactive Motion Technologies, Inc., Watertown, MA, USA) system has two translational degrees of freedom (dof): shoulder abduction-adduction (ab-ad), elbow flexion-extension (flexext).
  The robotic system supports the execution of reaching movements in the horizontal plane through an assist as needed control strategy. The robot can guide the movement of the upper limb of the patients and record end-effector physical quantities such as the position, velocity, and applied forces. The device is designed to have a low intrinsic end-point impedance (i.e., be back-drivable to easily carry the weight of the patient's arm, to execute movements without constraint and offer minimal resistance. A 3-dof force transducer is placed at the robots end-effector, as well.
  Other Names: MIT-MANUS/InMotion2
  Arms: Robot Group
Procedure: Traditional physiotherapy — Active or passive exercises.
  Other Names: FKT
  Arms: Traditional physiotherapy

SUMMARY:
Numerous studies showed that ascertaining the effectiveness of rehabilitative interventions on conditions leading to long-term disability, such as stroke, is a complex task because the outcome depends on many interacting factors. Several studies underline the importance of brain plasticity and its therapeutic potential in neurological disorders. Accredited theories of cortical reorganization after brain lesion endorse the use of early, intensive, repetitive, and context-related exercise as optimal strategies to promote motor relearning and minimize motor deficit. The use of robotic systems in upper limb motor rehabilitation programs has been already demonstrated to provide safe and intensive treatment to subjects with motor impairments due to a neurological injury: several studies showed the advantages of robotic therapy on chronic post-stroke patients, even if no consistent influence on functional abilities was found and evidence of better results providing intensive treatments, both robotic and conventional rehabilitative techniques, was found. Recent development and recent trial in robot-assisted rehabilitation has shown the great potential of robotic devices for delivering repetitive training, thus facilitating a high intensity and a large dose of training during sub-acute and chronic phases of stroke rehabilitation. The proposed project, through a randomized controlled observer-blind multicenter trial is aimed at evaluating the effectiveness of robot-assisted therapy as additional treatment to the standard physical therapy in the early phase after stroke onset and evaluating in conjunction with EEG and EMG recordings the effects of the rehabilitative treatments in a quantitative, measurable way, by providing reliable and objective methods for measuring functional recovery after stroke.

DETAILED DESCRIPTION:
The main original contribution of this project is to provide an experimental framework, based on proximal robotic treatment approach, to test whether starting with the distal robot-assisted sensorimotor therapy the effective in improving motor functions of sub-acute stroke patients.

The use of robotic platforms to administer the rehabilitation therapy is crucial for two main reasons:

1. the physical therapies based on robotic platforms assure that each patient in the same testing group is treated in the same repeatable way, eliminating the intrinsic subject-dependent variability that affects traditional therapies;
2. the robotic platforms, in conjunction with EEG and EMG recordings, can be used to assess the effects of the rehabilitative treatments in a quantitative, measurable way, by providing reliable and objective methods for measuring functional recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* first acute event of cerebrovascular stroke
* unilateral paresis,
* ability to understand and follow simple instructions,
* ability to remain in a sitting posture, even through seat belts for trunk fixation.

Exclusion Criteria:

* bilateral impairment,
* severe sensory deficits in the paretic upper limb,
* cognitive impairment or behavioral dysfunction that would influence the ability to comprehend or perform the experiment,
* refusal or inability to provide informed consent
* other current severe medical problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fugl-Meyer Scale at 28 weeks. | at inclusion, week 4 and week 28
Change from Baseline in Box and Block Test at 28 weeks. | at inclusion, week 4 and week 28.

SECONDARY OUTCOMES:
Change from Baseline in Modified Ashworth Scale at 28 weeks. | at inclusion, week 4 and week 28.

OTHER OUTCOMES:
Change from Baseline in Frenchay Arm Test at 28 weeks. | at inclusion, week 4 and week 28.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Goffredo, BME, Principal Investigator — IRCCS San Raffaele Rome
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Roma, Roma
  - Auxilium Viate Volterra, Volterra